CLINICAL TRIAL: NCT00539617
Title: A Single-Arm, Phase II Study of Tarceva Plus FOLFOX6 in Patients With Unresectable or Metastatic Cancer of Esophagus or Gastroesophageal Junction
Brief Title: Chemotherapy & Erlotinib in Treating Patients w/ Esophageal or Gastroesophageal Cancer That Cannot Be Removed by Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: For slow accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 064511; NCI-2011-01276 (Registry Identifier: NCI Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Esophageal Cancer
Keywords: metastatic esophageal cancer; erlotinib; folfox; advanced esophageal cancer; unresectable esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Erlotinib Hydrochloride; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tarceva and FOLFOX (Experimental): COMBINATION THERAPY PHASE: Patients receive erlotinib hydrochloride orally (PO) once daily (QD) on days 1-56. Patients also receive FOLFOX6 therapy comprising oxaliplatin intravenously (IV) over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46-48 hours on days 1, 15, 29, and 43. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity. Patients with stable disease or no evidence of disease after course 2 or subsequent courses continue on to maintenance phase.
  MAINTENANCE PHASE: Patients receive erlotinib hydrochloride PO QD on days 1-42. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib; Drug: 5-fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Erlotinib — Tarceva single agent therapy: 150 mg/day PO
  Other Names: Tarceva
Drug: 5-fluorouracil — 5-FU bolus: 400 mg/m2 IV once every 2 weeks for 16 weeks 5-FU infusion: 2400 mg/m2 IV over 46-48 hours, once every 2 weeks for 16 weeks
  Other Names: 5-FU; Adrucil
Drug: Leucovorin — 400 mg/m2 IV once every 2 weeks for 16 weeks
  Other Names: Folinic acid
Drug: Oxaliplatin — 85 mg/m2 IV once every 2 weeks for 16 weeks
  Other Names: Eloxatin

SUMMARY:
The purpose of this study is to test the safety and effectiveness of erlotinib and FOLFOX in patients with esophageal or gastro-esophageal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
More than 50% of patients with advanced esophageal cancer present with disease that cannot be removed by surgery or has spread to other parts of the body. Improved therapies for patients with advanced esophageal cancer are therefore urgently needed. The epidermal growth factor receptor (EGFR) inhibitor erlotinib (in combination with chemotherapy) has lead to improved survival in patients with pancreatic and lung cancer. EGFR is a target in esophageal cancer therapy since its overexpression is associated with more aggressive disease and poor survival. Early studies have shown some clinical activity of EGFR inhibitors in this disease alone or in combination with chemotherapy. This study aims to explore how safe and effective treatment with erlotinib and FOLFOX is in patients with advanced esophageal or gastro-esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal carcinoma (squamous or adenocarcinoma)
* Surgically unresectable disease and/or metastatic disease; endoscopic accessibility of the primary tumor is preferred but not a prerequisite
* No prior chemotherapy therapy except for neoadjuvant treatment (radiation and/or chemotherapy); prior treatment with EGFR-inhibiting agents is not allowed
* Life expectancy > 12 weeks
* Patients must have the ability to take and retain oral medications or have an appropriate percutaneous feeding tube in place
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (Karnofsky Performance Status (KPS) >= 50%)
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria and radiographic imaging performed within 28 days prior to registration
* Absolute neutrophil count (ANC) >= 1500/mL
* Platelet count >= 100,000/mL
* Hemoglobin level >= 10.0 gm/dL
* Serum creatinine =< 1.5 x IULN (institutional upper limits of normal); OR measured creatinine clearance >= 60 mL/min
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase (SGOT)) or alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase (SGPT)) =< 2.5 x IULN (unless the liver is involved by tumor, in which case it must be =< 5.0 x IULN)
* Total bilirubin =< 1.5 x IULN
* Provision of written informed consent
* Women of childbearing potential (WOCBP) must be willing to practice acceptable methods of birth control to prevent pregnancy; WOCBP are any females who have experienced menarche and who have not undergone surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), who are not postmenopausal (defined as amenorrhea >= 12 consecutive months), or are on hormone replacement therapy; acceptable methods of birth control include oral or hormonal contraceptives and barrier methods (e.g., condom, diaphragm) used in combination with other methods (e.g., spermicide)
* Male patients who are capable of fathering a child must avoid doing so while participating in this study through the use of acceptable methods of birth control; this is a precautionary measure because this study involves chemotherapy agents

Exclusion Criteria:

* Presence of a Kras mutation
* Lack of expression of EGFR (tumors that do not have detectable EGFR staining in at least 10% of tumor cells will not be considered EGFR-positive)
* Prior treatment with EGFR-inhibiting agents, chemotherapy, or radiotherapy for esophagogastric carcinomas (other than neoadjuvant treatment as noted in inclusion criteria)
* Patients must not be receiving any other investigational agents; use of erythropoietin is allowable; secondary prophylaxis with granulocyte colony stimulating factor (G-CSF) (Filgrastim) is allowable
* The patient concomitantly uses phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, or St. John's wort
* Uncontrolled brain metastases
* Patients must not have uncontrolled intercurrent illness at the time of registration including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina, pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not have current New York Heart Association Class III or IV heart disease
* Known human immunodeficiency virus (HIV) infection
* Pregnant or breast-feeding women
* Patients who have had prior malignancies, except non-melanoma skin cancer (basal or squamous cell carcinoma) are not eligible for this study; unless greater than 5 years has passed since the event
* Known severe hypersensitivity to Tarceva
* Treatment with a non-approved or investigational drug within 30 days before day 1 of trial treatment
* Incomplete healing from previous oncologic or other major surgery
* Serum creatinine level greater than Common Toxicity Criteria (CTC) grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-10-05 (Actual); Primary Completion 2011-05-12 (Actual); Study Completion 2011-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Michael Korn, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment is performed in the Helen Diller Family Comprehensive Cancer Center at University of California, San Francisco
Pre-assignment Details: This trial has a pre-enrollment phase in which patients have their tissue tested for Kras and EGFR mutations to determine eligibility for the treatment trial. There is also a run-in phase with Erlotinib followed by a post-treatment biopsy. After this, the main treatment phase begins.
Groups:
- FOLFOX and Erlotinib: Single arm study of FOLFOX6 plus Erlotinib
Period: Pre-screening Period
Arm/Group | FOLFOX and Erlotinib
Started | 7
Completed | 4
Not Completed | 3
Period: Run-In Period
Arm/Group | FOLFOX and Erlotinib
Started | 4
Completed | 3
Not Completed | 1
Period: Treatment Period
Arm/Group | FOLFOX and Erlotinib
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FOLFOX and Erlotinib
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from enrollment into the run-in period of the study to objective tumor progression as determined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria. The proportion of patients with PFS will be reported and evaluated using Kaplan-Meier survival curves with median survival and 95% confidence interval.
Time Frame: Up to 2 years
Population: No data was collected for progression free survival
Arm/Group | FOLFOX and Erlotinib
Number analyzed (Participants) | 0

2. Secondary Outcome: Objective Response Rate (RR)
Description: The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for Progressive Disease (PD) the smallest measurements recorded since the treatment started). Best response assignment will depend on the achievement of both measurement and confirmation criteria using RECIST for both target and non-target lesions. For target lesions, response is defined as follows: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): >= 30% decrease in sum of the LD, taking as reference the baseline sum LD; PD: >=20% increase in sum of the LD of target lesions, taking as reference smallest sum LD recorded since treatment started or appearance of one or more new lesions , Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: Up to 2 years
Population: No data was collected for overall response rate
Arm/Group | FOLFOX and Erlotinib
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Progression (TTP)
Description: Patient with objective tumor response or stable disease will be treated with single agent Tarceva until tumor progression. For this study, time to progression will be determined as the number of days following the first day of single agent treatment with Tarceva following the last and completed cycle of Tarcerva/FOLFOX combination therapy. TTP will be calculated for the entire patient population as well as for patients that objectively responded to the combination therapy versus those that did not.
Time Frame: Up to 2 years
Population: No data was collected for time to progression
Arm/Group | FOLFOX and Erlotinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Adverse events were collected from first dose to 30 days after last dose for the 4 patients who started treatment.
Arm/Group | FOLFOX and Erlotinib
All-Cause Mortality (participants affected / at risk) | 3/4
Serious Adverse Events (participants affected / at risk) | 4/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX and Erlotinib (N=4)
Dehydration (Gastrointestinal disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFOX and Erlotinib (N=4)
Abdomimal distention (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 3 (7)
Anorexia (Gastrointestinal disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema, limbs (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 4 (6)
Hypothroidism (Endocrine disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutrophil (Blood and lymphatic system disorders) | 3 (3)
Oral Pain (Gastrointestinal disorders) | 1 (1)
Pain, other (General disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Taste Alteration (Gastrointestinal disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight loss (General disorders) | 1 (1)
Tongue Ulcer (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to low accrual resulting in a sample size insufficient to conduct reliable analyses

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No